CLINICAL TRIAL: NCT01771133
Title: Pregnancy and EARly Lifestyle Improvement Study
Acronym: PEARLS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting or enrolling participants has halted prematurely by Life-Moms Consortium and will not resume; participants are no longer being examined or treated.
Sponsor: University of Puerto Rico (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kaumudi Joshipura, Director of the Center for Clinical Research and Health Promotion, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01HD072834 (NIH); U01HD072834 (NIH)
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Hyperglycemia
Keywords: Obesity; Maternal Welfare; Child Welfare; Nutritional Sciences; Clinical Trial; Pregnancy; Physical activity; Fetal Development; Metabolic Diseases; Life style; Behavior and Behavior Mechanisms; LIFE-Moms
MeSH Terms: conditions — Obesity; Hyperglycemia; Motor Activity; Metabolic Diseases; Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle and nutrition control group (No Intervention): The control arm will receive routine prenatal care in the prenatal clinic. They will receive regular phone calls and mailings, token gifts and some useful information from data collected in the study, such as physical activity, feedback on behavior throughout the study. To additionally promote adherence (since they will have less contact with study staff), we will include 2 pre-partum and 1 post-partum group sessions meant to increase bonding between participants and retention of control participants. These sessions will include general pregnancy information not related to our interventions.
- Lifestyle intervention group (Active Comparator): The lifestyle intervention will be delivered within an empowerment framework which promotes behavioral changes by facilitating health self-efficacy, utilizing self-praise and using active coping skills to address and manage emotions. A nutrition component primarily focuses on total calories, for which energy requirements will be individually calculated for each pregnant women and on general diet quality with an emphasis on carbohydrate quality. It will also promote an overall healthy diet, emphasizing improvement of fat quality and reducing salt intake. A physical activity component focuses on promoting regular movement and minimizes the duration of bouts of sitting or lying during waking hours as well as non-exercise activity.
  Interventions: Behavioral: Lifestyle intervention group

INTERVENTIONS:
Behavioral: Lifestyle intervention group — The lifestyle intervention will be delivered within an empowerment framework which promotes behavioral changes by facilitating health self-efficacy, utilizing self-praise and using active coping skills to address and manage emotions. A nutrition component primarily focuses on total calories, for which energy requirements will be individually calculated for each pregnant women and on general diet quality with an emphasis on carbohydrate quality. It will also promote an overall healthy diet, emphasizing improvement of fat quality and reducing salt intake. A physical activity component focuses on promoting regular movement and minimizes the duration of bouts of sitting or lying during waking hours as well as non-exercise activity.
  Arms: Lifestyle intervention group

SUMMARY:
The investigators propose to conduct a randomized controlled trial in 200 overweight/obese pregnant women and their offspring. The prenatal intervention will emphasize improving diet and physical activity. The lifestyle intervention will be delivered within an empowerment theoretical framework through a combination of group sessions, individual counseling, and by monitoring compliance to diet and physical activity to further tailor the intervention. The post-partum intervention sessions will include mothers and their offspring and will focus on breastfeeding, improving physical activity and quality of the diet and feeding practices through the first post-partum year. As part of routine prenatal care, participants in both the control and intervention arms will be given health-related advice. Since the majority of participants are expected to be eligible for the Women, Infants and Children (WIC) program, both groups will also receive assistance through WIC as per their routine policies. Our primary outcome is Gestational Weight Gain (GWG). The major secondary outcome of interest is infant BMI z-score at 12 months of age, and the investigators will also be evaluating several metabolic outcomes in mothers and infants.

DETAILED DESCRIPTION:
Obesity and hyperglycemia in pregnancy are thought to impact fetal growth through over-nutrition and may stress the fetal pancreas because of the increased demand for insulin. Such intrauterine programming events affect birth weight and raise the offspring's risk trajectory for future obesity, type 2 diabetes, cardiovascular disease and premature death. Investigators propose to conduct a randomized controlled trial in 200 overweight or obese pregnant Puerto Rican women (free of diabetes) and their infants, to favorably impact metabolic health in mothers and infants.

Women presenting will be randomized to a lifestyle modification intervention or standard care control group before 16 gestational weeks. The intervention will focus on improving: (1) physical activity levels and (2) diet quality and calorie intake. The lifestyle intervention will be delivered within an empowerment theoretical framework through individualized intervention sessions, intensive group sessions, and by phone calls. The intervention will continue through the first postpartum year and will include the infants. A key objective is to evaluate whether the intervention optimizes infant BMI z-score. We will also evaluate whether the intervention increases the number of women who experience appropriate gestational weight gain, and evaluate several additional aims including relating the interventions with improved insulin sensitivity and beta-cell function in the women, and insulin concentrations adjusted for glucose in their infants.This study will also help us to identify and overcome barriers to develop effective ways of intervening during pregnancy to meaningfully improve cardio-metabolic risk trajectories of future generations.

ELIGIBILITY:
Inclusion Criteria:

* Singleton viable pregnancy. A twin pregnancy reduced to singleton before 14 weeks by project gestational age is acceptable. An ultrasound must be conducted before randomization that shows a fetal heartbeat; there should be no evidence of more than one fetus on the most recent pre-randomization ultrasound.*
* Gestational age at randomization no earlier than 9 weeks 0 days and no later than 15 weeks 6 days based on an algorithm that compares the last menstrual period (LMP) date and data from the earliest ultrasound.*
* BMI ≥25 kg/m2 based on first trimester measured weight and on measured height. The earliest weight measurement before randomization, measured specifically for the study will be used. Reported pre-pregnancy weight will not be used to determine eligibility because of the potential for inaccuracy. If the earliest weight measurement is conducted at 140 to 146 weeks or 150 to 156 weeks, 1 lb or 2 lbs will be subtracted from the measured weight respectively, to adjust to a first trimester weight.*
* Age ≥ 18*

Exclusion Criteria:

* Diagnosis of diabetes prior to pregnancy (reported physician diagnosed diabetes other than GDM in previous pregnancy or taking insulin or medications to treat diabetes), or an HbA1c ≥ 6.5 % or other test result (elevated fasting glucose ≥126 mg/dL/7.0 mmol/L or 2 h glucose ≥200 mg/dL/11.1 mmol/L when OGTT is completed) suggestive of pre-pregnancy diabetes. All potential participants will have HbA1c performed prior to randomization.*
* Known fetal anomaly *
* Planned termination of pregnancy*
* History of three or more consecutive first trimester miscarriages*
* Past history of anorexia or bulimia by medical history or patient report. Binge eating disorder is not an exclusion*
* Current eating disorder diagnosed by EDE-Q questions 2-4 and confirmed after discussion with the participant by study staff*
* Actively suicidal defined as a value ≥ 2 on the BDI-II question 9*
* Prior or planned (within 1 year of expected delivery) bariatric surgery*
* Current use of one or more of the following medications: *

  * Metformin
  * Systemic steroids
  * Antipsychotic agents
  * Anti-seizure medications or mood stabilizers that would be expected to have a significant impact on body weight
  * Medications for ADHD including amphetamines and methylphenidate
* Continued use of weight loss medication including OTC and dietary supplements for weight loss *
* Contraindications to aerobic exercise in pregnancy specified in the ACOG Committee Opinion #267, 2002 (reaffirmed 2009) *

  * Hemodynamically significant heart disease defined as an AHA class II (short of breath with exercise) or greater
  * Restrictive lung disease (e.g. pulmonary fibrosis)
  * Poorly controlled seizure disorder
  * Poorly controlled hypertension (blood pressure ≥160/110)
  * History of extreme sedentary lifestyle (e.g. bed bound)
  * Orthopedic limitations to aerobic exercise
  * Severe anemia defined as a hemoglobin < 8 g/dl or hematocrit <24 %
* Participation in another interventional study that influences weight control*
* Enrollment in this trial in a previous pregnancy*
* Intention of the participant or of the care provider for the delivery to be outside the LIFE-Moms Consortium hospital*
* Participant's unwillingness or inability to commit to a 1 year follow-up of herself or her child, including planning to move away*
* Past or current intravenous drug use (visual check for injection marks, recorded methadone use, self-report)
* Self-reported HIV infection (confirmed from medical records or baseline test results)
* Inability to functionally participate in group sessions and other study requirements on a regular basis during the complete duration of the study, including but not limited to the documented use of the accelerometer for the periods required by the study
* Non Spanish speaking
* Plan on giving up infant for adoption

'*' Core eligibility criterion for the LIFE-Moms Consortium

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Gestational Weight Gain | Delivery
  To determine if a combined lifestyle intervention of nutrition and physical activity delivered within an empowerment theoretical framework in pregnant women result in a greater percent of women who gain the appropriate amount of gestational weight gain, as defined by the Institute of Medicine, compared to those receiving standard care.

SECONDARY OUTCOMES:
Does the lifestyle intervention (compared with control) affect the infant BMI z-score at 12 months of age (major | 12 months post-partum
  To evaluate whether the intervention influences infant BMI by comparison of infants of mothers randomized to either active intervention or control intervention
Estimates of beta-cell function and insulin action in the mother. | 35,0-36,6 wks 48,0-56,0 wks pp
  Estimation of beta-cell function, insulin resistance, and insulin sensitivity using data obtained from a frequently sampled 75g OGTT. Calculations will be based on established equations that have been validated for use in pregnancy, such as the model-based approach and the oral disposition index.
Maternal blood pressure during pregnancy | 24,0-27,6 wks; 35,0-36,6 wks; Delivery
Maternal blood pressure postpartum. | 4,0-6,0 wks pp; 16,0-24,0 wks pp; 48,0-56,0 wks pp
Infant blood pressure | < 48 hour pp; 4-6 wks pp; 16-24 wks pp
Post-partum weight retention | 4,0-6,0 wks pp; 16,0-24,0 wks pp; 48,0-56,0 wks pp
Body circumferences in mothers | 24,0-27,6 wks 35,0-36,6 wks 4,0-6,0 wks pp; 16,0-24,0 wks pp; 48,0-56,0 wks pp
Body circumferences in infants | < 48 hour pp 4-6 wks pp 16-24 wks pp 48-56 wks pp
Skinfold measures in infants | < 48 hour pp 16-24 wks pp 48-56 wks pp
Sleep quality and duration in the prenatal periods in mothers | 35,0-36,6 wks
  Sleep quality and duration will be assessed using an accelerometer in order to assess duration and quality of sleep
Sleep quality and duration in the postpartum periods in mothers and infants | 48,0-56,0 wks pp
  Sleep quality and duration will be assessed using an accelerometer in order to assess duration and quality of sleep
Insulin levels adjusted for glucose levels in the infants | < 48 hour pp 16-24 wks pp 48-56 wks pp
Developmental measures in infants | < 48 hour pp 16-24 wks pp 48-56 wks pp
Anthropometric and growth measures in the infants | < 48 hour pp 4-6 wks pp 16-24 wks pp 48-56 wks pp
Psychosocial measures in the mothers | 35,0-36,6 wks 48,0-56,0 wks pp
Pregnancy and Delivery complications | 35,0-36,6 wks delivery
Fetal and neonatal adverse outcomes | Birth and < 48 hour pp

OTHER OUTCOMES:
Additional Outcome Measures | 12 months
  Is there an interaction between gestational glucose abnormalities and physical activity/nutrition on infant outcomes?
Additional Outcome Measures | Pre-partum and post-partum
  What is the contribution of the different intervention components and varying levels of compliance on the maternal and infant outcomes as it is important to assess the feasibility of the intervention and the positive lifestyle changes in women and their infants assigned to the intervention compared to the control group?
Additional Outcome Measures | Pre-partum and post-partum
  Does the sleep quality and duration have an impact on glucose tolerance or GWG?
Additional Outcome Measure | Pregnancy
  GIS (Geographic Information Systems) will be used to evaluate the association between participants' environments in terms of proximity to parks and recreation facilities, restaurants, mass transit, etc and the major study outcomes, as well as compliance with physical activity and nutrition interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Kaumudi J Joshipura, ScD MS, Principal Investigator — University of Puerto Rico Medical Science Campus; Paul W Franks, PhD MPhil MS, Principal Investigator — Lund University
Locations (1):
- University of Puerto Rico Medical Science Campus, San Juan, Puerto Rico

REFERENCES:
- [Derived] Cabre HE, Drews KL, Pomeroy J, Keadle SK, Arteaga SS, Franks PW, Haire-Joshu D, Knowler WC, Pi-Sunyer X, Van Horn L, Wing RR, Cahill AG, Clifton RG, Couch KA, Gallager D, Josefson JL, Joshipura K, Klein S, Martin CK, Peaceman AM, Phelan S, Thom EA, Redman LM; LIFE-Moms Research Group. LIFE-Moms: effects of multicomponent lifestyle randomized control trial on physical activity during pregnancy in women with overweight and obesity. Int J Behav Nutr Phys Act. 2025 Sep 30;22(1):119. doi: 10.1186/s12966-025-01805-9. PMID 41029405
- [Derived] Flanagan EW, Drews KL, Cade WT, Franks PW, Gallagher D, Phelan S, Van Horn L, Redman LM. Metabolic Health and Heterogenous Outcomes of Prenatal Interventions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528264. doi: 10.1001/jamanetworkopen.2025.28264. PMID 40839263
- [Derived] Redman LM, Drews KL, Klein S, Horn LV, Wing RR, Pi-Sunyer X, Evans M, Joshipura K, Arteaga SS, Cahill AG, Clifton RG, Couch KA, Franks PW, Gallagher D, Haire-Joshu D, Martin CK, Peaceman AM, Phelan S, Thom EA, Yanovski SZ, Knowler WC; LIFE-Moms Research Group. Attenuated early pregnancy weight gain by prenatal lifestyle interventions does not prevent gestational diabetes in the LIFE-Moms consortium. Diabetes Res Clin Pract. 2021 Jan;171:108549. doi: 10.1016/j.diabres.2020.108549. Epub 2020 Nov 22. PMID 33238176
- [Derived] Peaceman AM, Clifton RG, Phelan S, Gallagher D, Evans M, Redman LM, Knowler WC, Joshipura K, Haire-Joshu D, Yanovski SZ, Couch KA, Drews KL, Franks PW, Klein S, Martin CK, Pi-Sunyer X, Thom EA, Van Horn L, Wing RR, Cahill AG; LIFE-Moms Research Group. Lifestyle Interventions Limit Gestational Weight Gain in Women with Overweight or Obesity: LIFE-Moms Prospective Meta-Analysis. Obesity (Silver Spring). 2018 Sep;26(9):1396-1404. doi: 10.1002/oby.22250. Epub 2018 Sep 6. PMID 30230252
- [Derived] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836